CLINICAL TRIAL: NCT03963440
Title: Cross-cultural Validation in French Language of the Questionnaire EARS Adapted to the Chronic Low Back Pain
Brief Title: Validation in French Language of the Questionnaire EARS
Acronym: EARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RNI 2018 COUDEYRE; 2018-A00616-49 (Other: 2018-A00616-49)
Record Dates: First submitted 2019-05-02; First posted 2019-05-24 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2019-05

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Physical activity; Questionnaire; Adhesion
MeSH Terms: conditions — Motor Activity; Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: Cross-cultural validation study of a questionnaire, interventional research involving the human person chronic low back pain, prospective, with cross-sectional cohort follow-up, multi-centric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohorte 1 (Experimental): Inclusion and first questionnaires period (10 questionnaires), after geting consent, during normal patient consultation schedule for functional restoration program of the lumbar spine (1 to 3 weeks hospital in day care).
  Second questionnaire period at 48h (Only EARS questionnaire) Third questionnaires period (10 questionnaires) at the end of the restoration program hospital care.
  Fourth and last questionnaires period (10 questionnaires) at 3 months during a normal patient follow-up consultation No additional appointments.
  Interventions: Other: Exercise Adherence Rating Scale (EARS)

INTERVENTIONS:
Other: Exercise Adherence Rating Scale (EARS) — Inclusion and first questionnaires period (10 questionnaires), after geting consent, during normal patient consultation schedule for functional restoration program of the lumbar spine (1 to 3 weeks hospital in day care).
  Second questionnaire period at 48h (Only EARS questionnaire) Third questionnaires period (10 questionnaires) at the end of the restoration program hospital care.
  Fourth and last questionnaires period (10 questionnaires) at 3 months during a normal patient follow-up consultation No additional appointments.
  Other Names: Quebec Back Pain Disability Scale; International Physical Activity Scale (IPAQ); Hospital Anxiety and Depression (HAD); Evaluation du fardeau lié à la réalisation des exercices physiques (ETBQ); Back Belief Questionnaire (BBQ); Arthritis Self-Efficacy Scale pour les lombalgies chroniques (ASES); Return To Work Self Efficacy Scale (RTWSE-10 items); Fear Avoidance Belief Questionnaire (FABQ); Impression globale de changement par le patient (PGIC)

SUMMARY:
The main objective of this work is to validate in French the questionnaire EARS, adapted to chronic low back pain.

Physical exercise is often recognized as necessary for primary and secondary prevention and treatment of chronic diseases. This is particularly true of chronic low back pain. It is therefore of paramount importance that compliance with such treatment be assessed to allow for readjustments, as well as drug treatment. No gold standard6-7 measured patient adherence to exercise programs until the creation of the EARS in 2016 by E.Godfrey and his team (Exercise Adherence Rating Scale, literally "joining physical exercise programs")

EARS is a reliable and validated psychometric assessment questionnaire that assesses adherence to prescribed physical exercise in chronic low back pain.

DETAILED DESCRIPTION:
Self-management of the patient to perform these exercises involves good collaboration with the care prescriber, leaving patients to manage and monitor their health. Long-term adherence to care programs, including physical exercise, is paramount for these patients in order to maintain a beneficial long-term effect, which is the case in non-specific chronic low back pain. However, evidence shows that compliance levels following a physical exercise prescription are low, limiting the benefits this could bring.

Currently, EARS is validated for chronic low back pain in its English version. To our knowledge and to the knowledge of the questionnaire's author, E.Godfrey, there are no other studies that have examined the validation of EARS in the French language for chronic low back pain.

Patients will be asked to complete a series of questionnaires after completing the non-opposition form. The management of non-specific chronic low back pain also requires evaluation through questionnaires, in accordance with the usual practices of the services participating in the study. No intervention will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Adult (>18 years old)
* Chronic Low Back Pain evolving for at least 3 months
* Acceptance to participate in the study
* Patients affiliated to a social security scheme (beneficiary entitled)

Exclusion Criteria:

* Patient under guardianship, or protection of justice.
* Patient in the incapacity to answer the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Psychometric properties of the French questionnaire EARS | 0 day, 2 days, 15 days, 3 months
  (acceptability, internal validity, reproducibility, convergent validity and validity of structure against external criteria)

SECONDARY OUTCOMES:
The fears and the faiths measured by questionnaire FABQ | at day 0, 15 days, 3 months
  The FABQ can help predict those that have a high pain avoidance behavior. Clinically, these people may need to be supervised more than those that confront their pain.
  The FABQ contains 2 scales: a work scale (FABQ-W) composed of 7 items and a physical activity scale (FABQ-PA) composed of 4 items. The two scales are scored separately. Higher FABQ scores indicate elevated fear-avoidance beliefs.
  "FABQ-W" has a point score that ranges from 0-42 points. It can be calculated as follows: (Total points for items 6, 7, 9, 10 11, 12 and 15) = Work scale score.
  "FABQ-PA" can range from 0-24 points. Scores are calculated as follows: (Total points for items 2, 3, 4 and 5) = Physical activity scale score.
The 14-item Beliefs and Behaviors Questionnaire (BBQ) measures beliefs, experiences and adherent behavior related with Low Back pain | at day 0, 15 days, 3 months
  The questionnaire consists of 14 items and each item is scored on a 5-point Likert agreement scale (ranging from strongly agree to strongly disagree). Only nine items are used in the scoring of the questionnaire with the remaining items considered 'distracters' from which no scores are derived. Possible scores range between 9 and 45, with lower scores indicating more maladaptive or pessimistic beliefs about back pain.
The knowledge of emotional state measured by questionnaire HAD | at day 0, 15 days, 3 months
  The Hospital Anxiety and Depression Scale (HADS) is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. HADS gives clinically meaningful results as a psychological screening tool and can assess the symptom severity and caseness of anxiety disorders and depression in patients with illness and the general population.
  One questionnaire, comprising fourteen questions. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  Scoring :
  0-7- normal, 8-10-borderling abnormal, 11-21-abnormal
Self-assessment of the incapacity, that deals with the echo on the everyday life measured by questionnaire QUEBEC | at day 0, 15 days, 3 months
  This questionnaire is about the way your back pain is affecting your daily life. People with back problems may find it difficult to perform some of their daily activities. For each activity there is a scale of 0 to 5 :0 - " not difficult at all " , 1 - " minimally difficult " , 2 - " somewhat difficult " , 3 - " fairly difficult " , 4 - " very difficult " and 5 - " unable to do ". Minimum detectable change (90% confidence) 15 points.
Evaluation of the burden, bound to the realization of the physical exercises by questionnaire ETBQ | at day 0, 15 days, 3 months
  (Exercise Therapy Burden Questionnaire), consisting of 10 items. For each activity there is a scale of 0 to 10 : 0 - not agree at all, 10 - completely agree. Some items of the ETBQ belong to side effects and others to the workload of health care. (lower score=better)
The personal efficacy by means of the questionnaire ASES "Arthritis Self-Efficacy Scale" | at day 0, 15 days, 3 months
  The ASES includes 20 questions that represent three subscales: pain, function, and other symptoms. Score ranging : from 1 to 10 (higher = greater self-efficacy).
The evaluation of the self-efficiency perceived of return in the work by means of the questionnaire RTWSE (10 items) | at day 0, 15 days, 3 months
  10-item RTWSE scale with the goal of assessing self-efficacy of workers to return to work within two conceptual domains: controlling pain at work and obtaining help. For each question there is a scale of to 5: 1 - not sure at all, 5 - really sure. Higher score = better self-efficiency.
Level of physical activity measured by short questionnaire IPAQ | at day 0, 15 days, 3 months
  Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). Scoring a HIGH level of physical activity on the IPAQ means your physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level Scoring a MODERATE level of physical activity on the IPAQ means some activity more than likely equivalent to half an hour of at least moderate intensity physical activity on most days.
  Scoring a LOW level of physical activity on the IPAQ means any of the criteria for either MODERATE of HIGH levels of physical activity.
Patient Global Impression of Change by Scale PGIC | 15 days, 3 months
  This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status. It consists of one item.
  Patient choose: 1 -No change (or condition has gotten worse), 2 - Almost the same, hardly any change at all, 3 - A little better, but no noticeable change, 4 - Somewhat better, but the change has not made any real difference, 5 - Moderately better, and a slight but noticeable change, 6 - Better and a definite improvement that has made a real and worthwhile difference, 7 - A great deal better and a considerable improvement that has made all the difference.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, MD-PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (5):
- France (5):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Lille, Lille
  - CHU de Montpellier, Montpellier
  - CHU de nîmes, Nîmes
  - Hôpital COCHIN, Paris

REFERENCES:
- [Background] Waddell G. 1987 Volvo award in clinical sciences. A new clinical model for the treatment of low-back pain. Spine (Phila Pa 1976). 1987 Sep;12(7):632-44. doi: 10.1097/00007632-198709000-00002. PMID 2961080
- [Background] Beinart NA, Goodchild CE, Weinman JA, Ayis S, Godfrey EL. Individual and intervention-related factors associated with adherence to home exercise in chronic low back pain: a systematic review. Spine J. 2013 Dec;13(12):1940-50. doi: 10.1016/j.spinee.2013.08.027. Epub 2013 Oct 26. PMID 24169445
- [Background] Bocerean C, Dupret E. A validation study of the Hospital Anxiety and Depression Scale (HADS) in a large sample of French employees. BMC Psychiatry. 2014 Dec 16;14:354. doi: 10.1186/s12888-014-0354-0. PMID 25511175
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Hall AM, Kamper SJ, Hernon M, Hughes K, Kelly G, Lonsdale C, Hurley DA, Ostelo R. Measurement tools for adherence to non-pharmacologic self-management treatment for chronic musculoskeletal conditions: a systematic review. Arch Phys Med Rehabil. 2015 Mar;96(3):552-62. doi: 10.1016/j.apmr.2014.07.405. Epub 2014 Aug 6. PMID 25108098